CLINICAL TRIAL: NCT05688995
Title: COVID-19 Vaccines and the Menstrual Cycle; a Cross-sectional Study
Brief Title: COVID-19 Vaccines and the Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Associate Professor, University of Jordan
Other Study IDs: ju
Record Dates: First submitted 2023-01-17; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Menstrual Irregularity
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Naser Al-Husban — COVID-19 vaccines

SUMMARY:
The study aimed to explore the effect of different COVID-19 vaccines on menstrual cycle

DETAILED DESCRIPTION:
This is a descriptive cross-sectional study that took place between September 2021 and December 2021. The study aimed to explore the effect of different COVID-19 vaccines on menstrual cycle. It used an anonymous questionnaire distributed via social media platforms; Facebook, Twitter, and WhatsApp across different cities of Jordan. A total of 732 responses were received with a 59% response rate.

The questionnaire was distributed over four months directed at women who have received at least one dose of the COVID-19 vaccine and who live in Jordan. It took 10 minutes to complete all the questions.

Data collection did not involve direct contact with participants to prevent the spread of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* less than 40 years
* healthy women
* received covid-19 vaccine

Exclusion Criteria:

* women who did not receive the vaccine
* those living outside Jordan (those cannot fill the form) and during analysis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with menstrual cycle
Study Population: Our study included 617 Menstruating females. 74.55% of participants were of the age group between 20-35 years. 59.64% had normal BMI (18.5-24.9 Kg/m2), while 11.99% were underweight (BMI less than 18.5 Kg/m2), 19.77% were overweight (BMI>24.9 Kg/m2 but less than 30 Kg/m2), and 8.59% were obese (BMI more than 30 Kg/m2). Largest BMI was 39.79 Kg/m2. Most of participants were single ladies (79.25%). 82.01% were nulliparous. 17.83% were multiparous, including 1.62% ladies that had 5 or more children (grand multiparous).
Sampling Method: Non-Probability Sample
Enrollment: 617 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
significant changes in the menstrual cycle after vaccination | 6 months
  changes that involve bleeding amount or pain

CONTACTS AND LOCATIONS:
Overall Officials: Naser U Al-Husban, Principal Investigator — The University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
can be shared with reasonable request from the primary investigator